CLINICAL TRIAL: NCT07381621
Title: A Prospective Evaluation of the Clinical Effectiveness of Perineural Dextrose and Conventional Local Anesthetic Injections in Patients With Symptomatic Knee Osteoarthritis
Brief Title: Perineural Dextrose Versus Local Anesthetic Injections in Knee Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nadide Koca, Principal Investigator, M.D., Physical Medicine and Rehabilitation, Ankara Training and Research Hospital
Other Study IDs: AnkaraTRH-FTR-NK-10; 2024-KAEK-40 (Other: Ankara Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Perineural Injection; Dextrose Injection; Local Anesthetic Injection; Pain; WOMAC; Observational Study
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perineural 5% Dextrose Group: Patients with symptomatic knee osteoarthritis receiving perineural 5% dextrose injections as part of routine clinical care.
  Interventions: Procedure: Perineural 5% Dextrose Injection
- Perineural Local Anesthetic Group: Patients with symptomatic knee osteoarthritis receiving perineural local anesthetic injections as part of routine clinical care.
  Interventions: Procedure: Perineural Local Anesthetic Injection

INTERVENTIONS:
Procedure: Perineural 5% Dextrose Injection — Perineural injection of 5% dextrose solution administered around periarticular sensory nerves of the knee as part of routine clinical practice.
  Groups: Perineural 5% Dextrose Group
Procedure: Perineural Local Anesthetic Injection — Perineural injection of local anesthetic administered around periarticular sensory nerves of the knee as part of routine clinical practice.
  Groups: Perineural Local Anesthetic Group

SUMMARY:
This prospective observational study aims to compare the clinical effectiveness of perineural 5% dextrose injections and perineural local anesthetic injections in patients with symptomatic knee osteoarthritis. Adult patients receiving routine perineural injection therapy will be followed for six months. Pain intensity and functional outcomes will be assessed at baseline and at 1, 3, and 6 months after treatment using validated clinical assessment tools.

DETAILED DESCRIPTION:
Knee osteoarthritis is a common degenerative joint disease associated with chronic pain, functional limitation, and reduced quality of life. Various non-surgical treatment modalities have been used to manage symptoms; however, the effectiveness of these treatments may be limited due to the complex pain mechanisms involved in osteoarthritis.

Perineural injection therapy has gained increasing attention as a minimally invasive treatment option targeting neurogenic inflammation around peripheral sensory nerves. Perineural 5% dextrose injection is thought to reduce pain by modulating neurogenic inflammation, while local anesthetic injections are commonly used in clinical practice for symptomatic relief.

This study is designed as a prospective observational cohort study conducted in a routine clinical setting. Patients aged 40 to 65 years with symptomatic knee osteoarthritis who are treated with perineural injections as part of standard care will be included. The choice of injectate (perineural 5% dextrose or perineural local anesthetic) will be determined based on clinical considerations and patient preference; no randomization or protocol-driven assignment will be performed.

Pain severity will be evaluated using the Visual Analog Scale (VAS). Functional status will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Additional clinical parameters, including knee range of motion measured by goniometry and quadriceps muscle strength assessed by manual muscle testing, will also be recorded. Assessments will be performed at baseline, and at 1, 3, and 6 months following treatment.

Clinical outcomes of the two treatment groups will be compared to evaluate changes in pain and functional status over time. The findings of this study are expected to contribute real-world evidence regarding the clinical effectiveness of perineural 5% dextrose and local anesthetic injections in the management of symptomatic knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis
* Clinical/radiological diagnosis
* Knee pain ≥ 3 months
* Written informed consent

Exclusion Criteria:

* Prior knee surgery
* Recent intra-articular injection
* Inflammatory rheumatic disease
* Severe systemic or neurological disease
* Pregnancy or breastfeeding

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 40 to 65 years with symptomatic knee osteoarthritis who are receiving perineural injection therapy as part of routine clinical care. Eligible participants include both male and female patients who meet the predefined inclusion and exclusion criteria and are able to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Intensity (Visual Analog Scale [VAS]) | Baseline, 1 month, 3 months, and 6 months
  Change in Knee Pain Intensity (Visual Analog Scale [VAS]) Change from baseline in knee pain intensity measured using the Visual Analog Scale (VAS), a 100-mm horizontal line anchored at 0 = no pain and 100 = worst imaginable pain; higher scores indicate worse pain.

SECONDARY OUTCOMES:
Change in Functional Status (Western Ontario and McMaster Universities Osteoarthritis Index [WOMAC]) | Baseline, 1 month, 3 months, and 6 months
  Change from baseline in WOMAC total score (and/or subscales: pain, stiffness, and physical function) assessing knee osteoarthritis-related symptoms. The WOMAC consists of 24 items with a total score ranging from 0 to 96; higher scores indicate worse symptoms and worse functional status.
Change in Knee Range of Motion | Baseline, 1 month, 3 months, and 6 months
  Change in knee joint range of motion measured using goniometry.
Change in Quadriceps Muscle Strength | Baseline, 1 month, 3 months, and 6 months
  Change in quadriceps muscle strength assessed by manual muscle testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital Ankara, Altindag, Turkey, 06230, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This is an observational, single-center study conducted in a hospital setting. The study includes sensitive clinical information, and individual-level data cannot be sufficiently de-identified for public sharing. Only aggregate results will be reported in scientific publications.

REFERENCES:
- [Background] Pan PJ, Wang JC, Tsai CC, Kuo HC. Identification of early response to hypertonic dextrose prolotherapy markers in knee osteoarthritis patients by an inflammation-related cytokine array. J Chin Med Assoc. 2022 Apr 1;85(4):525-531. doi: 10.1097/JCMA.0000000000000693. PMID 35019866
- [Background] Salsabil JR, Pane RV, Hasan H, Al Hajiri AZZ. Hypertonic Dextrose Prolotherapy Injection in Grade IV Knee Osteoarthritis with Obesity: A Case Report. Acta Med Indones. 2024 Jul;56(3):349-355. PMID 39463100
- [Background] Huang K, Cai H. Hypertonic dextrose prolotherapy in osteoarthritis: mechanisms, efficacy, and future research directions. Front Endocrinol (Lausanne). 2025 Aug 4;16:1602727. doi: 10.3389/fendo.2025.1602727. eCollection 2025. PMID 40831953
- [Background] Arias-Vazquez PI, Tovilla-Zarate CA, Legorreta-Ramirez BG, Burad Fonz W, Magana-Ricardez D, Gonzalez-Castro TB, Juarez-Rojop IE, Lopez-Narvaez ML. Prolotherapy for knee osteoarthritis using hypertonic dextrose vs other interventional treatments: systematic review of clinical trials. Adv Rheumatol. 2019 Aug 19;59(1):39. doi: 10.1186/s42358-019-0083-7. PMID 31426856
- [Background] Chen YW, Lin YN, Chen HC, Liou TH, Liao CD, Huang SW. Effectiveness, Compliance, and Safety of Dextrose Prolotherapy for Knee Osteoarthritis: A Meta-Analysis and Metaregression of Randomized Controlled Trials. Clin Rehabil. 2022 Jun;36(6):740-752. doi: 10.1177/02692155221086213. Epub 2022 Mar 8. PMID 35257594
- [Background] Bae G, Kim S, Lee S, Lee WY, Lim Y. Prolotherapy for the patients with chronic musculoskeletal pain: systematic review and meta-analysis. Anesth Pain Med (Seoul). 2021 Jan;16(1):81-95. doi: 10.17085/apm.20078. Epub 2020 Dec 16. PMID 33348947
- [Background] Hung CY, Hsiao MY, Chang KV, Han DS, Wang TG. Comparative effectiveness of dextrose prolotherapy versus control injections and exercise in the management of osteoarthritis pain: a systematic review and meta-analysis. J Pain Res. 2016 Oct 18;9:847-857. doi: 10.2147/JPR.S118669. eCollection 2016. PMID 27799816
- [Background] Jahangiri A, Moghaddam FR, Najafi S. Hypertonic dextrose versus corticosteroid local injection for the treatment of osteoarthritis in the first carpometacarpal joint: a double-blind randomized clinical trial. J Orthop Sci. 2014 Sep;19(5):737-43. doi: 10.1007/s00776-014-0587-2. Epub 2014 Aug 27. PMID 25158896
- [Background] Sit RWS, Wu RWK, Reeves KD, Rabago D, Chan DCC, Yip BHK, Chung VCH, Wong SYS. Efficacy of intra-articular hypertonic dextrose prolotherapy versus normal saline for knee osteoarthritis: a protocol for a triple-blinded randomized controlled trial. BMC Complement Altern Med. 2018 May 15;18(1):157. doi: 10.1186/s12906-018-2226-5. PMID 29764447
- [Background] Arden NK, Perry TA, Bannuru RR, Bruyere O, Cooper C, Haugen IK, Hochberg MC, McAlindon TE, Mobasheri A, Reginster JY. Non-surgical management of knee osteoarthritis: comparison of ESCEO and OARSI 2019 guidelines. Nat Rev Rheumatol. 2021 Jan;17(1):59-66. doi: 10.1038/s41584-020-00523-9. Epub 2020 Oct 28. PMID 33116279
- [Background] Fu Y, Du Y, Li J, Xi Y, Ji W, Li T. Demonstrating the effectiveness of intra-articular prolotherapy combined with peri-articular perineural injection in knee osteoarthritis: a randomized controlled trial. J Orthop Surg Res. 2024 May 5;19(1):279. doi: 10.1186/s13018-024-04762-4. PMID 38705988
- [Background] Wu YT, Chen YP, Lam KHS, Reeves KD, Lin JA, Kuo CY. Mechanism of Glucose Water as a Neural Injection: A Perspective on Neuroinflammation. Life (Basel). 2022 Jun 2;12(6):832. doi: 10.3390/life12060832. PMID 35743863
- [Background] Guzel I, Gul D, Akpancar S, Lyftogt J. Effectiveness of Perineural Injections Combined with Standard Postoperative Total Knee Arthroplasty Protocols in the Management of Chronic Postsurgical Pain After Total Knee Arthroplasty. Med Sci Monit. 2021 Feb 6;27:e928759. doi: 10.12659/MSM.928759. PMID 33547269
- [Background] Garcia-Triana SA, Toro-Sashida MF, Larios-Gonzalez XV, Fuentes-Orozco C, Mares-Pais R, Barbosa-Camacho FJ, Guzman-Ramirez BG, Pintor-Belmontes KJ, Rodriguez-Navarro D, Brancaccio-Perez IV, Esparza-Estrada I, Bernal-Hernandez A, Gonzalez-Ojeda A. The Benefit of Perineural Injection Treatment with Dextrose for Treatment of Chondromalacia Patella in Participants Receiving Home Physical Therapy: A Pilot Randomized Clinical Trial. J Altern Complement Med. 2021 Jan;27(1):38-44. doi: 10.1089/acm.2020.0287. Epub 2020 Nov 20. PMID 33217236
- [Background] Ebnerasooli S, Barghi A, Nasseri K, Moghimi N. Peri-articular Dextrose Prolotherapy: Investigating the Effect of Injection Site on Knee Osteoarthritis Pain: A Double-Blind, Randomized, Clinical Trial. Anesth Pain Med. 2024 Mar 27;14(2):e140966. doi: 10.5812/aapm-140966. eCollection 2024 Apr. PMID 39411379